CLINICAL TRIAL: NCT00306774
Title: Trial of Vitamin D to Reduce the Progression of Knee Osteoarthritis: A Double-Blind, Placebo-Controlled Once Daily Dosing Regimen
Brief Title: Vitamin D to Slow Progression of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AR051361 (NIH); R01AR051361 (NIH)
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; vitamin D; knee pain; cartilage loss; WOMAC; MRI; cartilage volume; OA; physical function; web-based; internet-based
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive vitamin D (cholecalciferol)
  Interventions: Dietary Supplement: Vitamin D (cholecalciferol)
- 2 (Placebo Comparator): Participants will receive a matched placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D (cholecalciferol) — 2,000 IU vitamin D capsule per day for 2 years
  Arms: 1
Dietary Supplement: Placebo — Placebo capsule per day for 2 years
  Arms: 2

SUMMARY:
Knee osteoarthritis (OA) is a common and disabling health problem in older adults and for which there is no cure. The purpose of this study is to determine the effects of vitamin D on knee OA symptoms and physical function in adults aged 45 years and older.

DETAILED DESCRIPTION:
Symptomatic knee OA is one of the most frequent causes of limitation in lower limb tasks, especially in the elderly. Knee OA causes 68 million lost work days per year. OA is the most frequent reason for joint replacement, at a cost of billions of dollars per year. There are currently no completely effective medical remedies for OA. Pharmaceutical companies are trying to develop drugs that will slow the disease progression of OA; however, such medications will be expensive to use in a population in which OA is common. There is evidence that vitamin D supplementation, a simple and much cheaper intervention, may prove useful in slowing the progression of OA. Even if only modestly effective, it could have considerable impact in terms of reducing the societal burden of OA. Therefore, in the interests of public health, the efficacy of vitamin D supplementation as a disease-modifying treatment for OA needs to be tested in a rigorous clinical trial. Disease modification trials for knee OA have been difficult in the past due to limitations of radiographic techniques. Fortunately, magnetic resonance imaging (MRI) has emerged as a valid, precise, and reproducible tool for the measurement of damage of cartilage and joint structures. The purpose of this study is to evaluate the effects of vitamin D on knee OA symptoms and physical function in older adults.

Patients with symptomatic knee OA will be randomly assigned to receive vitamin D at 2,000 International Units (IU) a day or placebo. Each participant will be in the study for about 2 years. During that time, there will be 9 scheduled study visits (screening, Months 0, 2, 4, 8, 12, 16, 20, and 24) and interim safety visits as needed. Measurements of vital signs, a knee exam, blood and urine collection, pill counts, and completion of questionnaires will occur at all visits. Participants' physical function will be assessed at study entry and Months 0, 12, and 24. MRI, bone density scanning, and an assessment by the study staff will occur at Months 0, 12, and 24. Knee x-rays will occur at study screening and Month 24.

ELIGIBILITY:
Inclusion Criteria:

* Chronic knee discomfort based on affirmative response to the question "During the past 12 months, have you had pain, aching, or stiffness in or around your knee(s) on most days for at least one month?"
* WOMAC pain subscale score of at least 1
* Tibiofemoral OA on posterior anterior (PA) weight-bearing semi-flexed knee radiographs with severity equivalent to Kellgren and Lawrence grade of at least 2
* Clinical examination confirming knee pain or discomfort referable to the knee joint
* Prepared to refrain from use of glucosamine, chondroitin, MSM, DMSO, and doxycycline
* Pass faintness of heart trial period

Exclusion Criteria:

* Serum 25(OH) vitamin D level greater than 80 ng/ml
* Use of glucosamine, chondroitin, or doxycycline within 3 months of random assignment
* Use of MSM, DMSO within 3 months of random assignment
* Use of vitamin D supplements such that the total daily dose is greater than 1,000 IU or a single source is greater than 800 IU
* Intra-articular joint injections (e.g., glucocorticoid or haluronic acid formulations, within 3 months of random assignment)
* Chronic glucocorticoid use
* Hypercalcemia (total serum calcium greater than 10.5 mg/dL)
* Hypercalcuria (spot urine calcium: creatinine ratio of 0.275 for women and 0.325 for men, corresponding to 24-hour calcium excretion of 0.30 and 0.35 g, respectively)
* Estimated GFR less than 30
* Hyperparathyroidism (PTH greater than 65 pg/mL)
* History of lymphoma or sarcoidosis
* Reiter's syndrome
* Psoriatic arthritis
* Rheumatoid arthritis
* Ankylosing spondylitis
* Currently on treatment for tuberculosis
* Malabsorption disorders (e.g., advance liver disease, chronic renal disease-stage 4 or 5, Crohn's disease, Whipple's disease, celiac sprue)
* Serious medical conditions or impairments that, in the view of the investigator, would obstruct study participation
* Pregnancy
* Plan to permanently relocate from the region during the trial period
* Planned knee or hip arthroplasty during the study period
* Any contra-indication to having an MRI scan

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2006-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cartilage volume loss (MRI) | 2 years
Knee symptoms (WOMAC questionnaire) | 2 years

SECONDARY OUTCOMES:
Physical function | 2 years
Quality of life | 2 years
Pathological (MRI) severity global score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E. McAlindon, MD, MPH, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Division of Rheumatology, Boston, Massachusetts, United States

REFERENCES:
- [Result] Wang, J., Nuite, M., Wheeler, L.M., Badiani, P., Joas, J., McAdams, E.L., Fletcher, J., LaValley, M.P., Dawson-Hughes, B., McAlindon, T.E. Low Vitamin D Levels are Associated with Greater Pain and Slow Walking Speed in Patients with Knee Osteoarthritis (KOA). ACR Abstract #199 Arthritis & Rheumatism. 2007;56: 9 (supplement): S124.
- [Result] Nuite, M., Wang, J., Wheeler, L.M., Fletcher, J., Badiani, P., McAdams, E.L., Joas, J., LaValley, M.P., Dawson-Hughes, B., McAlindon, T.E. Don't Always Believe What You Are Told: A comparison of Self-Reported with Measured Weight and Height. ARHP Abstract #2049 Arthritis & Rheumatism. 2007;56: 9 (supplement): S779.
- [Result] L. M. Wheeler, J. Wang, M. Nuite, J. Fletcher, P. Badiani, E. L. McAdams, J. P. Joas, M. P. LaValley, B. Dawson-Hughes, T. E. McAlindon. Report of Daily Vitamin D Supplement Use is No Guarantee of Protection Against Vitamin D Deficiency in Knee Osteoarthritis Patients. OARSI Abstract #248 Osteoarthritis and Cartilage. 2007. Vol. 15 (Supplement A)
- [Result] G.H. Lo, M.H. Smith, E.L. McAdams, K.A. Carr, M. Nuite, B. Dawson-Hughes, N. Palermo, T.E. McAlindon. Baseline Vitamin D Status is Predictive of Longitudinal Change in Tibial BMD in Knee Osteoarthritis (OA). ACR Abstract #193 Arthritis & Rheumatism. 2008.
- [Result] E.L. McAdams, G.H. Lo, L.L. Price, M.H. Smith, K.A. Carr, M. Nuite, J.P. Joas, T.E. McAlindon. Varus-Valgus Static Malalignment does Not Predict Changes in Physical Function over a 1-year Period in People with Knee Osteoarthritis (OA). ACR Abstract #194 Arthritis & Rheumatism. 2008.
- [Result] M.H. Smith, G.H. Lo, M. Nuite, E.L. McAdams, K.A. Carr, J.P. Joas, B. Dawson-Hughes, N. Palermo, T.E. McAlindon. Increased Medial Tibial Bone Mineral Density (BMD) is Associated with Deterioration in Walking Ability and Pain in Individuals with Knee Osteoarthritis (KOA). ACR Abstract #697 Arthritis & Rheumatism. 2008.
- [Result] Lo G.H., McAdams E., Smith M., Carr K., Nuite M., Dawson-Hughes B., Palermo N., McAlindon T.E. Tibial Plateau Proximal and Distal Bone Behave Similarly: Both Are Associated with Features of Knee Osteoarthritis (KOA). OARSI Abstract #137 Osteoarthritis and Cartilage. 2008. Vol. 16 (Supplement 4)
- [Result] Hansberry S., Lo G., Carr K., McAlindon T., Ward R., Nuite M., Schneider E. Comparing Quantitative v. Semi-Quantitative Analysis of Cartilage Degradation and Its Association with Knee Pain. Poster # 1072 from Transactions of the 55th Annual Meeting of the Orthopaedic Research Society (ORS), Las Vegas, Feb. 2009.
- [Result] Grace H. Lo, Timothy E. McAlindon, Kimberly A. Carr, Melanie A. Ripley, Melynn Nuite, William F. Harvey. Varus Thrust Is Associated with Pain in Knee Osteoarthritis. Arthritis and Rheumatism. 2009; 60:10(supplement) S310, Abstract #831
- [Result] W.F. Harvey, J.Y. Lee, K.A. Carr, M.A. Ripley, M. Nuite, T. E. McAlindon, G.H. Lo. Varus Thrust Is Associated with Cartilage Loss in Knee Osteoarthritis. Arthritis and Rheumatism. 2009; 60:10(supplement) S77, Abstract #211
- [Derived] McAlindon T, LaValley M, Schneider E, Nuite M, Lee JY, Price LL, Lo G, Dawson-Hughes B. Effect of vitamin D supplementation on progression of knee pain and cartilage volume loss in patients with symptomatic osteoarthritis: a randomized controlled trial. JAMA. 2013 Jan 9;309(2):155-62. doi: 10.1001/jama.2012.164487. PMID 23299607
- [Derived] Lo GH, Harvey WF, McAlindon TE. Associations of varus thrust and alignment with pain in knee osteoarthritis. Arthritis Rheum. 2012 Jul;64(7):2252-9. doi: 10.1002/art.34422. PMID 22307813